CLINICAL TRIAL: NCT02548182
Title: Enhancing Physical Activity and Weight Reduction Through Smartcare and Financial Incentives: A Pilot Randomized Controlled Trial
Brief Title: Enhancing Physical Activity and Weight Reduction Through Smartcare and Financial Incentives
Acronym: EPAWROSFI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2-1-002-12
Record Dates: First submitted 2015-09-07; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): A standardized education material on diet, exercise, and behavior modification were provided to all participants, and each participant received a one-to-one education on diet and exercise from a trained nurse for 5 minutes each session.
- smartcare (Active Comparator): Participants allocated to a smartcare arms received the Fit.life™ wireless physical activity tracker (Fit.life™, Suwon, Korea) that measures daily and weekly physical activity. It is convenient for data upload via Bluetooth on participant mobile phone or wirelessly via a personal computer, and has been validated for measurement of free-living physical activity in adults [REF]. Participants allocated to a smartcare arms were also provided a standardized education material on diet, exercise, and behavior modification.
  Interventions: Device: smartcare
- smartcare plus financial incentives (Active Comparator): Participants in the 'smartcare plus financial incentive' arms were told that they are entitled to receive financial incentives depending on their achievement of the physical activity and weight target, and the amount they ca expect .The investigators provide financial incentives classified as process-based incentive and outcome-based incentive in addition to smartcare group intervention. A smartphone application was customized for the use of the investigators' intervention, different for the 'smart care' group and 'smartcare plus financial incentive' group.
  Interventions: Device: smartcare; Other: financial incentives

INTERVENTIONS:
Device: smartcare — Fit.life™ wireless physical activity tracker can measure daily physical activity including activity strength and time. It was chosen for its small size, accuracy in the measurement of physical activity, and convenient data upload via Bluetooth on participant mobile phone or wirelessly via a personal computer. Fit.life™ wireless physical activity tracker has been validated for measurement of free-living physical activity in adults [REF]. A smartphone application was customized for the use of the investigators' intervention, different for the 'smart care' group and 'smartcare plus financial incentive' group. The version for the latter group included the feature for the monitoring and feedback of financial incentives.
  Other Names: Fit.life™ wireless physical activity tracker
  Arms: smartcare; smartcare plus financial incentives
Other: financial incentives — Financial incentives are provided in the form of process-based and outcome-based incentive.(maximum 320,000KRW) Process-based incentives were based on daily physical activity level. Participants in the 'smart care plus financial incentive' arms could earn incentives of up to 10,000 KRW per week according to the following schedule: 1,000 KRW if a participant reached target amount of physical activity in a day / An additional 3,000 KRW if a participant reached target amount of physical activity every day in a week. Outcome-based incentives were based on achievement of weight loss target at each visit. 50,000 KRW if a participant reached weight loss target of 3% from the baseline body weight at visit 2 (4 week)/ 50,000 KRW in weight loss target of 5% from the baseline body weight at visit 3 (8 week) / 100,000 KRW in weight loss target of 7% from the baseline body weight at final visit 4 (12 week)
  Arms: smartcare plus financial incentives

SUMMARY:
The investigators are planning to conduct a pilot RCT of young obese population to evaluate the effect of smartcare with or without financial incentives for 12 weeks. Participants will be randomly assigned to a three-arm of control, smartcare, and smartcare plus financial incentives group.

DETAILED DESCRIPTION:
To test the feasibility and potential impact of smartcare with or without financial incentives, the study employed a three-arm, open label randomized controlled trial design: control, smartcare, and smartcare plus financial incentives. The investigators hypothesized that the 'smartcare + financial incentive' arm will show the greatest change in outcomes, followed by the 'smartcare' only arm, and lastly the control arm. Specific aims of the study are as follows:

* To quantify the effectiveness of a 'smartcare' intervention to promote physical activity and reduce weight over a 12 week period.
* To quantify the incremental effectiveness of adding financial incentives to 'smartcare' intervention

ELIGIBILITY:
Inclusion Criteria:

1. male students aged between 19 to 45;
2. body mass index ≥ 27;
3. smartphone user (either Android or iPhone);
4. able and willing to attend a four pre-specified visit during the study period.

Exclusion Criteria:

1. any treatment involving pharmacotherapy, procedure, or surgery;
2. use of any activity tracker device during the last three months.
3. Those who answered positively to any Physical Activity Readiness Questionnaire (PAR-Q) question were also excluded.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the amount of weight loss (kg) | 12 weeks
  Body weight change from the baseline body weight at each visit (4, 8, 12 week)

SECONDARY OUTCOMES:
the level of physical activity (METs*hour/week) | 12 weeks
  Average weekly physical activity(METs*hour/week) calculated by the IPAQ(International Physical Activity Questionnaire) at visit 4 (12 week), Physical activity change (METs*hour/week) from the baseline body weight at visit 4 (12 week)

CONTACTS AND LOCATIONS:
Overall Officials: Belong Cho, MD, MPH, PhD, Principal Investigator — Depart. of Family Medicine/Center for Health Promotion and Optimal Aging, Seoul National University Hospital

REFERENCES:
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Brennan TA, Asch DA, Volpp KG. Randomized trial of four financial-incentive programs for smoking cessation. N Engl J Med. 2015 May 28;372(22):2108-17. doi: 10.1056/NEJMoa1414293. Epub 2015 May 13. PMID 25970009
- [Background] Finkelstein EA, Linnan LA, Tate DF, Birken BE. A pilot study testing the effect of different levels of financial incentives on weight loss among overweight employees. J Occup Environ Med. 2007 Sep;49(9):981-9. doi: 10.1097/JOM.0b013e31813c6dcb. PMID 17848854
- [Background] Giles EL, Robalino S, McColl E, Sniehotta FF, Adams J. The effectiveness of financial incentives for health behaviour change: systematic review and meta-analysis. PLoS One. 2014 Mar 11;9(3):e90347. doi: 10.1371/journal.pone.0090347. eCollection 2014. PMID 24618584
- [Derived] Shin DW, Yun JM, Shin JH, Kwon H, Min HY, Joh HK, Chung WJ, Park JH, Jung KT, Cho B. Enhancing physical activity and reducing obesity through smartcare and financial incentives: A pilot randomized trial. Obesity (Silver Spring). 2017 Feb;25(2):302-310. doi: 10.1002/oby.21731. Epub 2017 Jan 7. PMID 28063226